CLINICAL TRIAL: NCT06235762
Title: Nutritional Intervention, Glycemic Control and Cardiovascular Outcomes in Participants With Type 2 Diabetes Mellitus
Brief Title: The Effects of Nutritional Intervention on Health Parameters in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Tatiana Palotta Minari, Principal Investigator, Sao Jose do Rio Preto Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33554520.0.0000.5415
Record Dates: First submitted 2023-12-22; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus Type 2; Diabetes Mellitus Type 2 in Obese; Diabetes; Diabetes Mellitus Non-insulin-dependent; Hypertension; Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Nutritional intervention; Nutrition; Nutritional Strategy; COVID-19; Mediterranean Diet; DASH Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension; COVID-19

STUDY DESIGN:
Intervention Model Description: Ranzomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Medical Evaluation (No Intervention): Participants in the control group will only undergo conventional medical evaluation.
- Conventional Medical Evaluation Plus Nutritional Assessment (Active Comparator): Participants in the intervention group will undergo the same medical care, concomitantly with nutritional assessment.
  Interventions: Behavioral: Nutritional Intervention

INTERVENTIONS:
Behavioral: Nutritional Intervention — This clinical trial evaluate the effects of nutritional intervention (individualized and personalized for each patient) on anthropometric, biochemical and cardiovascular parameters in participants with type 2 diabetes mellitus
  Arms: Conventional Medical Evaluation Plus Nutritional Assessment

SUMMARY:
The goal of this clinical trial is to evaluate the effects of nutritional intervention on anthropometric, biochemical and cardiovascular parameters in participants with type 2 diabetes mellitus. Participants will be distributed into 2 groups (control and intervention). Participants in the control group will only undergo conventional medical assessment and participants in the intervention group will receive the same medical care, concomitantly with nutritional assessment. The nutritional intervention is expected to reduce anthropometric data, glycemic and cardiovascular parameters in participants with T2DM, as opposed to the control group.

DETAILED DESCRIPTION:
The goal of this clinical trial is: 1- Evaluate the effects of nutritional intervention on anthropometric parameters {Weight, Body Mass Index (BMI), Waist Circumference and Waist Hip Ratio (WHR)}, biochemical parameters {Fasting blood glucose, Glycated Hemoglobin (HBA1C), Total Cholesterol ( TC), LDL Cholesterol (LDL-C), HDL Cholesterol (HDL-C) and Triglycerides} and cardiovascular {Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Heart Rate (HR)}. 2- Evaluate behavioral patterns related to lifestyle, such as skipping breakfast, sleep quality (induction, maintenance and awakenings) and frequency of physical activity. 3-Support knowledge to the participant to build eating autonomy, consequently improving quality of life in the long term.

This research will recruit participants diagnosed with T2DM (of both sexes aged between 18 and 80 years), at the Diabetes Outpatient Clinic and Hypertension at the Faculty of Medicine of São José do Rio Preto. The interventions will be distributed in quarterly meetings. Participants will be randomly distributed into 2 groups (control and the intervention group). The 40 participants in the control group will only undergo conventional medical evaluation and the 40 Participants in the intervention group will undergo the same medical care, concomitantly with nutritional assessment. Nutritional services will be made up of: A) Application of protocols (1-Nutritional History - Anthropometric, Biochemical and Clinical; 2-Habitual Food Record; 3-Sociodemographic protocol); B) Delivery of nutritional guidelines; C) Preparation of an individualized eating plan (inspired by the Mediterranean Diet and DASH diet with moderate carbohydrate content and restriction of saturated fats).

It is expected that interventions modulate the recovery of nutritional status, dietary inadequacies, parameters anthropometric, biochemical, cardiovascular and clinics, thus improving quality of life and reducing the risk of events in participants with T2DM in long term. In this way, the participants in treatment with nutritional support will be able to achieve greater benefit, maximizing the construction of a process of autonomy to feed.

ELIGIBILITY:
* Inclusion criteria - Participants with:

  * Age: Adults above 18 years to below 80 years.
  * Diagnosis of the disease: T2DM, that is, fasting blood glucose values equal to or greater than 126 mg/dL and glycated hemoglobin equal to or greater than 6.5%.
  * Gender: Male and female
  * Availability to participate in quarterly meetings during a period of 36 months.
  * Nutritional status: initial diagnosis of overweight or obesity, that is, with BMI above 24.9kg/m².
  * Sedentary.
* Exclusion criteria - Participants who:

  * They had difficulties answering the requested instruments.
  * They demonstrated impediments to assiduity in data collection.
  * They did not present a diagnosis of T2DM.
  * They were using insulin therapy.
  * They were using SGLT-2 inhibitors and/or GLP-1 analogues.
  * People with Chronic Kidney Disease.
  * Eutrophic or malnourished.
  * Physical exercisers, that is, more than 150 minutes of moderate to intense exercise per week.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-08-16 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | 12 months
  Evaluate the impact of nutritional intervention on weight (kg) between the 0th and 12th month.
Body Mass Index (kg/m²). | 12 months
  Evaluate the impact of nutritional intervention on Body Mass Index (kg/m²) between the 0th and 12th month.
Waist circumference (cm) | 12 months
  Evaluate the impact of nutritional intervention on Waist circumference (cm) between the 0th and 12th month.
Waist Hip Ratio (WHR) [Waist circumference (cm)/hip circumference(cm)] | 12 months
  Evaluate the impact of nutritional intervention on Waist Hip Ratio (WHR) between the 0th and 12th month.
fasting blood glucose concentration (mg/dl) | 12 months
  Evaluate the impact of nutritional intervention on Fasting blood glucose (mg/dl) between the 0th and 12th month.
glycated hemoglobin (HBA1C) rates (%) | 12 months
  Evaluate the impact of nutritional intervention on Glycated Hemoglobin (HBA1C) (%) between the 0th and 12th month.
Total Cholesterol ( TC) concentration (mg/dl) | 12 months
  Evaluate the impact of nutritional intervention on Total Cholesterol ( TC) (mg/dl) between the 0th and 12th month.
LDL Cholesterol (LDL-C) concentration (mg/dl) | 12 months
  Evaluate the impact of nutritional intervention on LDL Cholesterol (LDL-C) (mg/dl) between the 0th and 12th month.
HDL Cholesterol (HDL-C) concentration (mg/dl) | 12 months
  Evaluate the impact of nutritional intervention on HDL Cholesterol (HDL-C)(mg/dl) between the 0th and 12th month.
Triglycerides concentration (mg/dl) | 12 months
  Evaluate the impact of nutritional intervention on Triglycerides(mg/dl) between the 0th and 12th month.
Systolic Blood Pressure (SBP) (mmHg) | 12 months
  Evaluate the impact of nutritional intervention on Systolic Blood Pressure (SBP) (mmHg) between the 0th and 12th month.
Diastolic Blood Pressure (DBP) (mmHg) | 12 months
  Evaluate the impact of nutritional intervention on Diastolic Blood Pressure (DBP) (mmHg) between the 0th and 12th month.
Heart Rate (HR) beats per minute (bpm) | 12 months
  Evaluate the impact of nutritional intervention on Diastolic Blood Pressure (DBP) (mmHg) between the 0th and 12th month.

SECONDARY OUTCOMES:
Skipping breakfast (yes or no) | 12 months
  Observe changes in breakfast skipping habits between the 0th and 12th month.This qualitative variation will be measured by the standard protocol of conventional clinical nutritional analysis, using the metric of (yes or no). Individuals who report "yes" will be considered to have skipped breakfast and individuals who report "no" will be considered to have not skipped breakfast.
Sleep duration (hours) (more than 6 hours or less than 6 hours) | 12 months
  Observe changes in sleep duration (h) between the 0th and 12th month. This qualitative variation will be measured by the standard protocol of conventional clinical nutritional analysis, using the metric of (more than 6h or less than 6h of sleep). Individuals who report ">6" will be considered to have slept more than 6 hours per night and individuals who report "<6" will be considered to have slept less than 6 hours per night.
Night awakenings (amount/ number) | 12 months
  Observe changes in night awakenings between the 0th and 12th month. This qualitative variation will be measured by the standard protocol of conventional clinical nutritional analysis, using the metric of (more than 1 nighttime awakening or no nighttime awakenings). Individuals who report ">1" will be considered to have 1 or more awakenings and individuals who report "0" will be considered to have not awakened during sleep.
Physical activity level (sedentary, moderate, advanced) | 12 months
  Observe changes in Physical activity level between the 0th and 12th month. The presence or absence of physical exercise will be assessed through nutritional history. Patients with levels equal to or greater than 5 training sessions per week, with a total duration of 250 minutes/week, were considered very active/advanced. Patients with levels equal to or greater than 3 training sessions per week, with a total duration of 150 minutes/week, were considered active/moderate. Individuals below this recommendation were considered sedentary.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Palotta Minari, PhD Student, Principal Investigator — State Faculty of Medicine in São José do Rio Preto
Locations (1):
- Faculty of Medicine in São José do Rio Preto, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in nutritional strategies for the management of type 2 diabetes mellitus. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact:
  tatianaminari@gmail.com